CLINICAL TRIAL: NCT01291277
Title: Appropriate Time Interval for Repeat Sessions of Endoscopic Ligation for the Eradication of Esophageal Varices
Brief Title: Time Interval for Endoscopic Variceal Ligation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Yale University (Other); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Loren Laine, Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-08-00172
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Variceal Bleeding
Keywords: gastrointestinal hemorrhage; esophageal varices; gastrointestinal endoscopy; ligation
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ligation: 1-week interval (Active Comparator): Endoscopic variceal ligation performed at 1-week intervals
  Interventions: Device: Endoscopic Variceal Ligation
- Ligation 2-week interval (Active Comparator): Endoscopic variceal ligation performed at 2-week intervals
  Interventions: Device: Endoscopic Variceal Ligation

INTERVENTIONS:
Device: Endoscopic Variceal Ligation — Ligation of esophageal varices
  Other Names: variceal banding

SUMMARY:
Patients with liver disease frequently present to the hospital with bleeding from dilated veins in their foodpipe (called esophageal varices). The current standard of care is to perform endoscopic variceal ligation (placing rubber bands around the varices through an endoscope)in patients presenting with bleeding varices. Patients generally receive ligation at the time they come in with bleeding and then return at regular intervals to have repeat ligation in order to eradicate the varices. However there have been no studies to determine the appropriate intervals for esophageal variceal ligation until eradication. We will conduct a randomized comparison of 1-week vs. 2-week intervals for esophageal ligation in patients that have presented with bleeding varices. Our hypothesis is that one-week ligation will achieve more rapid eradication than the two-week interval with a greater proportion of patients achieving variceal eradication at 4 weeks after the index bleeding episode.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with acute upper GI bleeding due to esophageal varices and underwent successful endoscopic variceal ligation.
* Patients who would normally receive repeat endoscopic ligation therapy to eradicate varices.

Exclusion Criteria:

* Persistent bleeding despite endoscopic and medical therapy
* Platelet count < 40,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-08; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, M.D., Principal Investigator — University of Southern California
Locations (1):
- L.A. County + U.S.C. Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ligation: 1-week Interval | Ligation 2-week Interval
Started | 45 | 45
Completed | 40 | 42
Not Completed | 5 | 3
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligation: 1-week Interval | Ligation 2-week Interval | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 66] | 54 [30 to 78] | 54 [27 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 31 | 38 | 69

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Eradication of Esophageal Varices
Time Frame: At 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ligation: 1-week Interval | Ligation 2-week Interval
Number analyzed (Participants) | 45 | 45
Participants | 37 | 23

ADVERSE EVENTS:
Arm/Group | Ligation: 1-week Interval | Ligation 2-week Interval
Serious Adverse Events (participants affected / at risk) | 16/45 | 15/45
Other Adverse Events (participants affected / at risk) | 4/45 | 1/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligation: 1-week Interval (N=45) | Ligation 2-week Interval (N=45)
Hospitalization (General disorders) | 16 | 15 — Per the study design, this predefined outcome that we collected and reported was the serious adverse event of hospitalization (not specific etiologies).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligation: 1-week Interval (N=45) | Ligation 2-week Interval (N=45)
Esophageal (Gastrointestinal disorders) | 4 | 1 — This predefined outcome included any of the esophageal symptoms of dysphagia, odynophagia, and/or chest pain (a composite endpoint).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No